CLINICAL TRIAL: NCT03165591
Title: Open Label Phase II Immunotherapy Trial of Inoperable Pancreatic Cancer
Brief Title: Open Label Immunotherapy Trial of Inoperable Pancreatic Cancer
Acronym: V3-P
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Immunitor LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Panc-001
Record Dates: First submitted 2017-05-18; First posted 2017-05-24 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Pancreatic Cancer Non-resectable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Daily tablet of V3-P given orally for 2 months
  Interventions: Biological: V3-P

INTERVENTIONS:
Biological: V3-P — one tablet of V3-P given once daily for 2 months
  Other Names: oral tableted therapeutic vaccine

SUMMARY:
Pancreatic cancer (PDA) is the most lethal form of cancer, and the fourth-leading cause of cancer-related death in the United States, with a survival rate of less than 7%.There are currently no treatments found to be effective for patients with advanced disease who are ineligible for surgery, a prognosis representing the majority of pancreatic cancer diagnoses. Pancreatic cancer is not amenable to chemotherapy as compared to other cancer types, leaving patients with practically no options except surgery.

We have made oral tableted therapeutic vaccine, V3-P, derived from pooled blood of patients with PDA in line with similar highly promising approach we have adopted for patients with hepatocellular carcinoma (HCC) and cholangiocarcinoma (CAA). Patients with PDA will be given one tablet per day of V3-P and followed up to see the outcome.

DETAILED DESCRIPTION:
This study is an open label Phase II study aimed to recruit at least 20 patients with inoperable PDA and who are positive for CA19.9 pancreatic tumor marker. The presence of higher than normal levels of CA19.9 is the sole inclusion criteria. Patients will be given one tablet of V3-P daily and followed for three months.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of inoperable pancreatic cancer
* higher than normal of serum CA19.9 tumor marker levels (40 IU/ml)
* must be able to swallow tablets

Exclusion Criteria:

* negative for CA19.9
* pregnant, breast feeding women
* unwillingness to provide written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect of V3-P on tumor burden | 3 months
  Changes in CA19.9 tumor marker induced by daily dose of oral vaccine V3-P in an open label trial in patients with inoperable pancreatic cancer.

SECONDARY OUTCOMES:
Safety of V3-P | 3 months
  Toxicity or adverse side effects, such as diarrhea and vomiting, will be graded according to accepted standards, e.g., NCI CTEP CTCAE.
Effect of V3-P on sugar and bilirubin levels | 3 months
  Monthly evaluation of fasting glucose and bilirubin levels as a surrogate for pancreatic function

CONTACTS AND LOCATIONS:
Overall Officials: Allen Bain, PhD, Study Chair — Immunitor Inc.
Locations (2):
- Mongolia (2):
  - Immunitor LLC, Ulaanbaatar
  - National Cancer Center, Ulaanbaatar

IPD SHARING:
Plan to Share IPD: Undecided
The data will be shared with other researchers upon request on study conclusion

REFERENCES:
- [Background] Tarakanovskaya MG, Chinburen J, Batchuluun P, Munkhzaya C, Purevsuren G, Dandii D, Hulan T, Oyungerel D, Kutsyna GA, Reid AA, Borisova V, Bain AI, Jirathitikal V, Bourinbaiar AS. Open-label Phase II clinical trial in 75 patients with advanced hepatocellular carcinoma receiving daily dose of tableted liver cancer vaccine, hepcortespenlisimut-L. J Hepatocell Carcinoma. 2017 Apr 12;4:59-69. doi: 10.2147/JHC.S122507. eCollection 2017. PMID 28443252